CLINICAL TRIAL: NCT05056298
Title: Effect of Adding Arch Support Insole to Foot Strengthening Exercise in Patients With Bilateral Flexible Flatfoot
Brief Title: Effect of Insole Added to Exercise in Patients With Bilateral Flexible Flatfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohamed Ramadan Ibraheem Ramadan, Principal investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ramadan_MSc
Record Dates: First submitted 2021-09-18; First posted 2021-09-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-09

CONDITIONS: Flat Feet; Flexible Flatfoot; Balance; Distorted; Muscle Weakness
MeSH Terms: conditions — Flatfoot; Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insole and Exercise group (Experimental): will contain 17 patients, they will receive the custom made arch support insole in addition to the strengthening of foot muscles both intrinsic and extrinsic muscles.
  Interventions: Other: Custom made insole; Other: Strengthening exercises of extrinsic foot muscles; Other: Strengthening exercises of intrinsic foot muscles
- Exercise group (Active Comparator): will contain 17 patients, they will receive the standard insole in addition to the strengthening of foot muscles both intrinsic and extrinsic muscles.
  Interventions: Other: Strengthening exercises of extrinsic foot muscles; Other: Strengthening exercises of intrinsic foot muscles; Other: Standard insole

INTERVENTIONS:
Other: Custom made insole — Custom made arch support insole with semi-rigid arch support will be made using the casting method, plaster cast of both feet in a subtalar neutral position will be taken from each subject by highly specialized orthotist. The negative casts will be placed in calcaneal vertical position and custommolded orthosis will be fabricated to positive molds obtained from the negative casts with the goal to control the pronation movement of the foot
  Arms: Insole and Exercise group
Other: Strengthening exercises of extrinsic foot muscles — Participants will perform extrinsic foot muscles strengthening exercises with both ankles 3 times per week, 20 minutes for 8 weeks. they will be trained using a progressive resistance protocol using Thera-Band elasticated bands. Subjects will be progressed weekly throughout the training period according to progressive resistance protocol for dorsiflexors, planterflexors, evertors and investors muscles.
Other: Strengthening exercises of intrinsic foot muscles — The patient will assume the same position as in intrinsic foot muscle assessment, then he will be instructed to hold the position for a count of 10 seconds and attempt to maintain the MLA as steady as possible during the entire time without any compensatory extrinsic foot muscle activity. Following the 10-seconds, slowly and with eccentric control allow the foot to pronate and the MLA to lower to a relaxed state .
Other: Standard insole — Patient will be instructed to wear a standard prefabricated flat insole as a placepo treatment iniside his shoes for 2 months (8 weeks), 6 to 8 hours per day, and adhere to wearing the orthoses during outdoor walking and during extrinsic foot muscle training.
  Arms: Exercise group

SUMMARY:
Pesplanus, commonly known as 'flatfoot,' is a common pathomechanical condition characterized by a lowered medial longitudinal arch (MLA) and exaggerated pronation. There are two general types of flatfoot : flexible flatfoot and rigid flatfoot Flexible flatfoot is the most common form of flat foot. In adult population, it was reported that prevalence of flexible flatfeet is 13.6%. It has been proved that there is static and dynamic balance deficit in the participants with flatfeet. The extrinsic muscles as posterior tibialis (TP) ) and intrinsic muscles as abductor hallucis (AbdH) act as active subsystem support for the MLA during weight-bearing, standing, and walking. Abnormal alignment of the foot may cause stretch weakness of the foot muscles by elongating beyond the neutral physiological resting position. leading to musculoskeletal dysfunction and overuse injuries. Insoles can assist in maintaining normal alignment of the foot, improve balance as it supports MLA which is essential to stabilize postural sway, they widen the contact surface of the sole of the foot improving stability.

DETAILED DESCRIPTION:
Insoles have been used to correct pathomechanical alterations that occur in patients with flexible flat feet, it was reported that they reduced ankle eversion, ankle inversion moment and reduced the load placed on the ankle invertor muscles which must act eccentrically to control over-pronation and support the arch. Insole with intrinsic foot muscle training has been reported to increase strength on flexor hallucis and cross-sectional area of the AbdH muscle in patient with pes planus. Therefore insole combined with short foot exercises is recommended for strengthening intrinsic foot muscles in pes planus.

Wearing hard insole has been reported to improve postural stability as it limits and control the range of foot pronation, correct foot malalignment and promotes a neutral foot position.

Many studies had investigated the effect of using insole alone or exercise program alone or comparing between them on flexible flat foot patients. Up to the knowledge of the primary investigator, this is the first study to investigate the effect of adding arch support insole to strengthening exercise of foot muscles (intrinsic or extrinsic) in terms of dynamic balance, foot function, and foot muscle strength (intrinsic or extrinsic).

ELIGIBILITY:
Inclusion Criteria:

1. Navicular drop tests (NDT) 10 mm or larger difference in the navicular tuberosity heights.
2. Age range from 18-30 years from both sexes to limit the effects of arthritic changes that would be caused by bilateral FFF over the age 30.
3. BMI 18-30 as the prevalence of flexible flatfoot appears to be higher in individuals with a higher body mass index (BMI).

Exclusion Criteria:

1. history of lower extremity injuries as fractures, congenital deformities or surgery affecting balance.
2. history of cerebral concussions affecting balance.
3. visual or vestibular disorders, and/or any neurological deficit affecting balance.
4. any sign of foot pain, history of patellofemoral pain syndrome, plantar fasciitis, TA or TP dysfunction affecting foot function and balance.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | at baseline and after 2 months of intervention
  assessing the change in dynamic balance via using star excursion balance test. The individual will be instructed to establish a stable base of support on the stance limb in the middle of the testing grid and maintain it through a maximal reach excursion in one of the prescribed directions. While standing on a single limb, the participant is asked to reach as far as possible with the reaching limb along each reaching line ; lightly touches the line with the most distal portion of the reaching foot without shifting weight to or coming to rest on this foot of the reaching limb, and the maximum reaching distance will be measured by tape measurement, then the participant is asked to return the reaching limb to the beginning position in the center of the grid, reassuming a bilateral stance.
Foot function | at baseline and after 2 months of intervention
  assessing the change in Foot function via using The arabic version of Foot and ankle ability measure questionnaire. It is a 29-item questionnaire divided into two subscales: the FAAM, 21-item Activities of Daily Living Subscale and the FAAM, 8-item Sports Subscale. • Scoring of each item will be based on a 5-point Likert scale (4 to 0) from no difficulty at all' to unable to do. Item score totals range from 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale. Higher scores represent higher levels of function for each subscale with 100% representing no dysfunction. The score on each of the items is added together to get the item score total which is divided by the highest potential score. This value is then multiplied by 100 to get a percentage
Extrinsic foot muscle strength | at baseline and after 2 months of intervention
  assessing the change in Extrinsic foot muscle strength via using Hand held dynamometer device. Participants will be placed in subtalar neutral position for all testing. The lower leg will be strapped down to stabilize and prevent any accessory movement. Participants will be instructed to pull or push against the device as hard as they could for each direction and the investigator will counteracte that force with both hands for 3 seconds per trial, 3 consecutive trials will be conducted with a 10-second rest between trials. The maximum force (newtons) was used for analysis as the patient peak force .
Intrinsic foot muscle strength | at baseline and after 2 months of intervention. • The therapist will Count to 30 seconds and will observe for the steadiness of the navicular height and for any compensatory extrinsic foot muscle activity
  assessing the change in Intrinsic foot muscle strength via using intrinsic foot muscle test.patient will be directed to Stand in front of a wall, with the feet shoulder width apart and knees slightly flexed. The fingertips may be lightly placed on the wall. In order to achieve subtalar joint neutral, the therapist will gently supinate the feet by lifting all the toes off the floor, then slowly drop the toes down again but maintain the MLA. This most often results in arise of the MLA and the navicular bone, due to the windlass effect via the plantar fascia. If this procedure proves difficult, then simply the patient will be ordered to increase the height of the MLA, by actively trying to approximate the head of the first metatarsal towards the heel, without flexing the toes. While maintaining the MLA, the patient will stand on a single leg, as steady as possible. The fingertips should remain lightly on the wall for balance and fall prevention

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ramadan, Demonstrator, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Horus University, Egypt, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No